CLINICAL TRIAL: NCT02299830
Title: Prospective, Open, Multicenter Study of Interventional Pulmonologic Treatment of Malignant Central Airway Stricture
Brief Title: Study of Interventional Pulmonologic Treatment of Malignant Central Airway Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: Changhai Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Xinqiao Hospital of Chongqing (Other); China Meitan General Hospital (Other); Micro-Tech (Nanjing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAO-NO.201402024-malignant1; NO.201402024 (Other Grant/Funding Number: National Health and Family Planning Commission)
Record Dates: First submitted 2014-10-26; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Airway Obstruction
Keywords: neoplasm; central airway; obstruction
MeSH Terms: conditions — Airway Obstruction; Neoplasms; Bites and Stings | interventions — Cryotherapy; Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- cryotherapy (Experimental): give the cases whose central airway stricture were caused by soft neoplasm tissues cryotherapy
  Interventions: Procedure: cryotherapy
- argon plasma coagulation (Experimental): give the cases whose central airway stricture were caused by hard neoplasm tissues argon plasma coagulation
  Interventions: Procedure: argon plasma coagulation
- stent (Experimental): give the cases whose central airway stricture were caused by neoplasm compression stent placement
  Interventions: Procedure: stent placement
- snare (Experimental): give the cases whose central airway stricture were caused by polypoid neoplasm tissues snare
  Interventions: Procedure: deletion tumor tissue by snare

INTERVENTIONS:
Procedure: cryotherapy — use cryotherapy to delete soft neoplasm tissue in the airway
  Arms: cryotherapy
Procedure: argon plasma coagulation — use argon plasma coagulation to delete hard neoplasm tissue in the airway
  Arms: argon plasma coagulation
Procedure: stent placement — use stent placement to open the airway compressed by out neoplasm
  Arms: stent
Procedure: deletion tumor tissue by snare — use snare to delete polypoid neoplasm tissue in the airway
  Arms: snare

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of four interventional pulmonology techniques for the treatment of malignant central airway stricture.

The four techniques are：

* cryotherapy
* argon plasma coagulation
* stent
* snare

ELIGIBILITY:
Inclusion Criteria:

* malignant neoplasm caused central airway stenosis
* the degree of stenosis is above 50%
* estimated survival duration is longer than 3 months
* received no treatment one month before
* can understand the statement informed consent
* agree to enroll in the study

Exclusion Criteria:

* older than 70 years or younger than 18 years
* not malignant neoplasm caused central airway stenosis
* not central airway stenosis
* existence of lumina collapse or twisting
* severe arrhythmia, myocardial ischemia or hypertensive crisis
* coagulation disorders
* existence of severe organ disfunction
* allergic to anesthesia drugs
* refuse to participate the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
percentage of the cases that got Ⅰand Ⅱlevel remission | the next day after the treatment

SECONDARY OUTCOMES:
the values of dyspnea index | the next day after the treatment
Karnofsky Physical scales | the next day after the treatment

OTHER OUTCOMES:
adverse event during the treatment | from the beginning of the treatment to 48 hours after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Faguang Jin, Ph.D, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China